CLINICAL TRIAL: NCT05406115
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 786 in Healthy Subjects and Subjects With Obesity
Brief Title: Single and Multiple Ascending Dose Study to Evaluate AMG 786 in Healthy Participants and Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20210011
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: Obesity; AMG 786; Metabolic Indication
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Single Ascending Dose Cohorts (Experimental): Participants in 4 cohorts will receive either AMG 786 or placebo in Single Ascending Doses.
  Interventions: Drug: AMG 786; Other: Placebo
- Part A: Food Effect Cohort (Experimental): Participants in the food effect cohort (FEC) will receive 1 of 2 AMG 786 in 1 of two sequences. Participants in Sequence 1 will receive a dose of AMG 786 on day 1 under fed conditions followed by a 10-day washout period and another dose of AMG 786 on day 11 under fasted conditions. Participants in Sequence 2 in the FEC cohort will receive the first dose on day 1 under fasted conditions and the second dose on day 11 under fed conditions.
  Interventions: Drug: AMG 786; Other: Placebo
- Part B: Multiple Ascending Dose Cohorts (Experimental): Participants in 4 cohorts will receive either AMG 786 or placebo in Multiple Ascending Doses.
  Interventions: Drug: AMG 786; Other: Placebo

INTERVENTIONS:
Drug: AMG 786 — Oral tablet
Other: Placebo — Oral tablet

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of AMG 786 as single or multiple doses in healthy and obese participants.

DETAILED DESCRIPTION:
The 4th Multiple Ascending Dose cohort was not started.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study-specific activities/procedures
* Age 18 to 65 years at the time of signing the informed consent
* Female participants must be of non-childbearing potential (as described below)

  * Postmenopausal is defined as:
* Age of ≥ 55 years with no menses for at least 12 months; OR
* Age < 55 years with no menses for at least 12 months AND with a follicle-stimulating hormone (FSH) level > 40 IU/L or according to the definition of "postmenopausal range" for the laboratory involved; OR
* History of hysterectomy; OR
* History of bilateral oophorectomy
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and Electrocardiograms (ECGs) on day -1 (Part A) and day -1 (Part B) and screening
* Body Mass Index must be between 18 and < 25 kg/m^2 for healthy participants and between ≥ 25 and ≤ 32.0 kg/m^2 for otherwise healthy participants with obesity
* Have a stable body weight (less than 5 kg self-reported change during the previous 8 weeks) prior to screening
* Willing to maintain current general diet and physical activity regimen, except for the physical activity in the 72 hours before each blood sample collection for the clinical laboratory analysis, which should not be strenuous

Exclusion Criteria:

* Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years
* History or clinical evidence of diabetes mellitus, including a fasting glucose ≥ 125 mg/dl (6.9 mmol/L) and/or HbA1c ≥ 6.5%
* Triglycerides ≥ 5.65 mmol/L (ie, 500 mg/dL) at screening
* Hepatic liver enzymes alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or total bilirubin levels > 1.5 times the upper limit of normal (ULN) at screening. Participants with suspected or diagnosed Gilbert's disease will be excluded from the study.
* History or clinical evidence of bleeding diathesis or any coagulation disorder, including prothrombin time (PT), activated partial thromboplastin time (APTT), International normalized ratio (INR) or platelet count outside of the laboratory's normal reference range unless interpreted as not clinically significant by the investigator in consultation with the medical monitor at screening.
* History of gastrointestinal (GI) abnormality that could affect GI motility (including small bowel or colonic resection, inflammatory bowel disease, irritable bowel disease, and colon or GI tract cancer)
* Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid-stimulating hormone (TSH) value outside normal range
* A corrected QT interval at screening of > 450 msec in males or > 470 msec in females or history of long QT syndrome
* History of coronary artery disease or congestive heart failure
* Participants with a history of renal impairment or renal disease and/or estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73 m^2
* Obesity induced by other endocrinologic disorders (eg, Cushing's Syndrome)
* Previous surgical treatment for obesity (excluding liposuction if performed > 1 year before trial entry)
* History of major depressive disorder
* History of other severe psychiatric disorders, eg, schizophrenia, bipolar disorder
* A patient health questionnaire-9 score of ≥ 10
* Participant has a history or evidence of suicidal ideation (severity of 3, 4 or 5) or any suicidal behavior based on an assessment with the Columbia suicide severity rating scale at screening
* Surgery scheduled for the trial duration period, except for minor surgical procedures, with consultation by the Amgen Medical Monitor
* Positive results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus ribonucleic acid (RNA). For hepatitis C, hepatitis C antibody (HepCAb) testing is done at screening, followed by hepatitis C virus RNA by polymerase chain reaction (PCR) if hepatitis C antibody is positive
* Participant has systolic blood pressure ≥ 150 mm Hg or diastolic blood pressure ≥ 90 mm Hg at screening, and on day -1. For each visit, if the initial blood pressure is elevated, the reading may be repeated once at least 15 minutes later and the lower of the 2 readings may be used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 through end of study (approximately 40 days)
  Any clinically significant changes in vital signs, 12-lead electrocardiograms (ECGs) and clinical laboratory tests will be recorded as TEAEs.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of AMG 786 | Day 1 through end of study (approximately 40 days)
Time of Maximum Observed Concentration (Tmax) of AMG 786 | Day 1 through end of study (approximately 40 days)
Area Under the Concentration-time Curve (AUC) of AMG 786 | Day 1 through end of study (approximately 40 days)
Cmax of Metabolite M5 | Day 1 through end of study (approximately 40 days)
Tmax of Metabolite M5 | Day 1 through end of study (approximately 40 days)
AUC of Metabolite M5 | Day 1 through end of study (approximately 40 days)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Translational Clinical Research LLC, Aventura, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com